CLINICAL TRIAL: NCT01058551
Title: Incidence of New Onset Atrial Fibrillation in Patients With Severe Obstructive Sleep Apnea: The Reveal XT-SA Study
Brief Title: Incidence of Atrial Fibrillation in Patients With Severe Obstructive Sleep Apnea: The Reveal XT-SA Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Adrian Baranchuk (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor-Investigator, Dr. Adrian Baranchuk, MD, Queen's University
Organization: Queen's University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Reveal XT-SA
Record Dates: First submitted 2010-01-27; First posted 2010-01-28 (Estimated); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Obstructive Sleep Apnea; Atrial Fibrillation
Keywords: Sleep Apnea; Atrial Fibrillation
MeSH Terms: conditions — Sleep Apnea, Obstructive; Atrial Fibrillation; Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Reveal XT ILR (Experimental): Implantable Loop Recorder Insertion
  Interventions: Device: Implantable Loop Recorder Insertion

INTERVENTIONS:
Device: Implantable Loop Recorder Insertion — Implantable Loop Recorder Insertion. The device will be explanted after reaching outcome (First AF detected) or at 36 months
  Other Names: Reveal XT ILR, Medtronic

SUMMARY:
Single site study: The goal of the study is to determine the incidence of new onset atrial fibrillation (AF) in patients with severe obstructive sleep apnea (OSA) syndrome through the use of a Medtronic Reveal XT implantable Loop recorder (ILR). The ILR device is approved for use in Canada, for the assessment of atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with severe OSA defined as Apnea Hypopnea Index (AHI) > 30.
2. Age > 18 years.

Exclusion Criteria:

1. Previous history of clinical AF defined as documented lone, paroxysmal, persistent or permanent, according to standard definitions.
2. Patient with anticipated requirement of MRI.
3. Patient with well-know allergy to any component of the Medtronic Reveal XT.
4. Patients with implantable cardiac rhythm device [pacemakers or internal cardiac device (ICDs)].
5. Women of child bearing potential.
6. Unable or unwilling to provide written informed consent.
7. Unable or unwilling to complete the study follow-up schedule (eg. intention to leave the Kingston area over the next 3 years.
8. Previously enrolled in this trial.
9. Enrolled in another study that would confound the results of this trial.
10. Documented history of heart failure
11. Diagnosed with severe obstructive sleep apnea greater than 1 year from screening date

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2011-06; Primary Completion 2019-09-10 (Actual); Study Completion 2019-09-18 (Actual)

PRIMARY OUTCOMES:
To determine the incidence of new onset AF in patient's with severe OSA | 36 months

SECONDARY OUTCOMES:
To determine the impact of continuous positive airway pressure (CPAP) treatment in patients with new onset of AF in patients with severe OSA. (post hoc analysis) | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Baranchuk, MD, Principal Investigator — Queen's University
Locations (1):
- Kingston General Hospital, Kingston, Ontario, Canada

REFERENCES:
- [Background] Baranchuk A, Simpson CS, Redfearn DP, Fitzpatrick M. It's time to wake up! Sleep apnea and cardiac arrhythmias. Europace. 2008 Jun;10(6):666-7. doi: 10.1093/europace/eun078. Epub 2008 Apr 7. No abstract available. PMID 18390984
- [Background] Kanagala R, Murali NS, Friedman PA, Ammash NM, Gersh BJ, Ballman KV, Shamsuzzaman AS, Somers VK. Obstructive sleep apnea and the recurrence of atrial fibrillation. Circulation. 2003 May 27;107(20):2589-94. doi: 10.1161/01.CIR.0000068337.25994.21. Epub 2003 May 12. PMID 12743002
- [Background] Gami AS, Pressman G, Caples SM, Kanagala R, Gard JJ, Davison DE, Malouf JF, Ammash NM, Friedman PA, Somers VK. Association of atrial fibrillation and obstructive sleep apnea. Circulation. 2004 Jul 27;110(4):364-7. doi: 10.1161/01.CIR.0000136587.68725.8E. Epub 2004 Jul 12. PMID 15249509
- [Derived] Yeung C, Drew D, Hammond S, Hopman WM, Redfearn D, Simpson C, Abdollah H, Baranchuk A. Extended Cardiac Monitoring in Patients With Severe Sleep Apnea and No History of Atrial Fibrillation (The Reveal XT-SA Study). Am J Cardiol. 2018 Dec 1;122(11):1885-1889. doi: 10.1016/j.amjcard.2018.08.032. Epub 2018 Sep 7. PMID 30274768